CLINICAL TRIAL: NCT01282437
Title: Prophylactic Cranial Irradiation (PCI) Versus Observation in Radically Treated Patients With Stage III Non-small Cell Lung Cancer; A Phase III Randomized Study.
Brief Title: Prophylactic Cranial Irradiation (PCI) vs Observation in Stage III NSCLC
Acronym: NVALT11
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: University Medical Center Groningen (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVALT11
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Non Small Cell Lung Cancer (NSCLC); Radical Treatment; Stage III Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylactic Cranial Irradiation (Experimental)
  Interventions: Radiation: Prophylactic Cranial Irradiation
- Observation (No Intervention): Patients will not receive PCI, but will be observed and the same items will be measured as in the PCI-arm.

INTERVENTIONS:
Radiation: Prophylactic Cranial Irradiation — * 18 fractions of 2Gy
  * 12 fractions of 2.5Gy
  * 10 fractions of 3 Gy
  Arms: Prophylactic Cranial Irradiation

SUMMARY:
For patients with stage III non-small cell lung cancer, which is radically treated, we will investigate whether prophylactic cranial irradiation (PCI) should become standard of care to prevent brain metastases.

DETAILED DESCRIPTION:
For this group of patients, brain metastases are one of the major sites of tumor failure. Radical therapy of symptomatic brain metastases is seldom possible and only very rarely, long term survival can be achieved. PCI has shown to reduce the incidence of brain metastases in patients with non-small cell lung cancer to the same extent as in limited disease small-cell lung cancer. However, the exact value of PCI in stage III NSCLC patient, treated with contemporary chemo-radiation schedule with or without surgery, remains unsettled. Therefore this study is launched, in order to investigate whether PCI should become the standard of care in patients with stage III NSCLC who are treated with curative intention.

ELIGIBILITY:
Inclusion Criteria:

* UICC stage IIIA or IIIB (without malignant pleural of pericardial effusion) non-small cell lung cancer (histology or cytology)
* Whole body FDG-PET-scan before start of therapy available: No distant metastases
* CT or MRI of the brain before the start of radical therapy available: No brain metastases
* Platinum-based chemotherapy is mandatory
* Radical local therapy: concurrent of sequential chemotherapy (platinum-based) and radiotherapy with or without surgery
* Radiotherapy dose without surgery at least a biological equivalent of 60Gy
* No prior cranial irradiation
* Patients must sign a study-specific informed consent at the time of registration

Exclusion Criteria:

* The opposite of the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2009-01; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients developing symptomatic brain metastasis | 24 months after randomisation

SECONDARY OUTCOMES:
Time to develop neurological symptoms (confirmed or unconfirmed by imaging) | 24 months after randomisation
Measurement of side effects (CTCAE3.0) | 24 months after randomisation
Quality of Life | 24 months after randomisation
  Measured by QLQ-C30 and EuroQol 5D

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD, PhD, Principal Investigator — NVALT oncology foundation; Harry Groen, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (9):
- Netherlands (9):
  - VU Medical Center, Amsterdam, Amsterdam
  - Maastro Clinic, Maastricht, Limburg
  - UMCG Groningen, Groningen, Provincie Groningen
  - UMC Utrecht, Utrecht, Utrecht
  - The Netherlands Cancer Institute, Amsterdam
  - RT Insitute Stedendriehoek, Deventer
  - St. Antonius Ziekenhuis, Nieuwegein
  - Dr. Bernard Verbeeten Institute, Tilburg
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] Witlox WJA, Ramaekers BLT, Joore MA, Dingemans AC, Praag J, Belderbos J, Tissing-Tan C, Herder G, Haitjema T, Ubbels JF, Lagerwaard J, El Sharouni SY, Stigt JA, Smit EF, van Tinteren H, van der Noort V, Groen HJM, De Ruysscher DKM. Health-related quality of life after prophylactic cranial irradiation for stage III non-small cell lung cancer patients: Results from the NVALT-11/DLCRG-02 phase III study. Radiother Oncol. 2020 Mar;144:65-71. doi: 10.1016/j.radonc.2019.10.016. Epub 2019 Nov 14. PMID 31733490